CLINICAL TRIAL: NCT01993758
Title: The Efficacy of Using Lower Tourniquet Pressure During Total Knee Arthroplasty: Comparison With Conventional Tourniquet Pressure Group
Brief Title: Efficacy of Lower Tourniquet Pressure During Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B-1310/221-007
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Osteoarthritis
Keywords: tourniquet pressure; total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional tourniquet pressure (Active Comparator): The patients in this group will undertake total knee arthroplasty under conventional tourniquet pressure, which will be set as the pressure added by 150mmHg on the last systolic blood pressure just before tourniquet inflation.
  Interventions: Procedure: Conventional tourniquet pressure
- Low tourniquet pressure (Experimental): The patients in this group will undertake total knee arthroplasty under low tourniquet pressure, which will be set as the pressure added by 120mmHg on the last systolic blood pressure just before tourniquet inflation.
  Interventions: Procedure: Low tourniquet pressure

INTERVENTIONS:
Procedure: Low tourniquet pressure — Tourniquet pressure set as 120mmHg above the systolic blood pressure just before tourniquet inflation
  Arms: Low tourniquet pressure
Procedure: Conventional tourniquet pressure — Tourniquet pressure set as 150mmHg above the systolic blood pressure just before tourniquet inflation
  Arms: Conventional tourniquet pressure

SUMMARY:
This study aims to determine whether the lower tourniquet pressure, which is set by adding 120mmHg (millimeter of mercury) on the systolic blood pressure just before tourniquet inflation, are efficient and safe during total knee arthroplasty, compared with the conventional tourniquet pressure: 150mmHg above the systolic blood pressure before tourniquet inflation.

DETAILED DESCRIPTION:
We will compare the two groups of patients undergoing total knee arthroplasty, which the tourniquet pressure will be set differently: systolic blood pressure plus 120mmHg vs. systolic blood pressure plus 150mmHg, the conventional method, in terms of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* The patients undergoing total knee arthroplasty

Exclusion Criteria:

* Systolic blood pressure measured at ward > 200mmHg
* Thigh circumference > 78cm
* Anesthesia other than spinal anesthesia
* Simultaneous bilateral total knee arthroplasty
* The patients who disagreed the enrollment of this study

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Acquisition of bloodless surgical field just after skin incision | just after skin incision during operation
  Dichotomous variable determined during operation by operator (Yes or No)

SECONDARY OUTCOMES:
Failure of acquiring bloodless surgical field during operation | after skin incision through the point of tourniquet deflation
Increasement of tourniquet pressure to acquire bloodless surgical field | after skin incision though the point of tourniquet deflation
  We will increase the tourniquet pressure by 30mmHg from the initial tourniquet pressure, if we will fail to achieve bloodless surgical field during operation. The increasement of tourniquet pressure will be recorded if it will be needed during operation.
Thigh pain on the site of tourniquet application | postoperative 2nd day
  measured by 11-point numerical visual analog scale (VAS)and 5-Likert scale
Knee pain | postoperative 2nd day
  measured by 11-point numerical visual analog scale (VAS)and 5-Likert scale
Skin problem on the site of tourniquet application | posteoperative 2nd day
  It includes ecchymosis, bullae formation and skin necrosis.
Nerve palsy | within 7 days after surgery
symptomatic venous-thromboembolism | within 7 days after surgery
  It includes deep vein thrombosis and pulmonary embolism which are symptomatic and diagnosed by confirmative test, such as CT angiogram.

CONTACTS AND LOCATIONS:
Overall Officials: T K Kim, MD, PhD, Principal Investigator — Joint Reconstruction Center, Seoul National University Bundang Hospital
Locations (1):
- Joint Reconstruction Center, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim TK, Bamne AB, Sim JA, Park JH, Na YG. Is lower tourniquet pressure during total knee arthroplasty effective? A prospective randomized controlled trial. BMC Musculoskelet Disord. 2019 Jun 4;20(1):275. doi: 10.1186/s12891-019-2636-7. PMID 31159799